CLINICAL TRIAL: NCT01063309
Title: Non-Invasive Assessment of Atherosclerosis in Patients With CGD and Other Disorders of the Immune System
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100029; 10-I-0029
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Atherosclerosis; Chronic Granulomatous Disease (CGD)
Keywords: CAT SCAN; Heart Disease; Magnetic Resonance Imaging; Electrocardiogram; Superoxide
MeSH Terms: conditions — Atherosclerosis; Granulomatous Disease, Chronic; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (7):
- Autosomal recessive CGD: Participants must have autosomal recessive CGD (p47phox, p67phox, or p22phox deficiency) as demonstrated by DHR or genetic screening.
- CGD carrier: Participants with confirmed as X-linked CGD carriers as demonstrated by DHR or genetic screening.
- Healthy Volunteer: Healthy volunteers over the age of 18, both male and female. That have not been diagnosed with CGD, Inflammatory Bowel Disease, or another primary disease of the immune system.
- IFN-gamma treated CGD: Participants with CGD the have been treated with Interferon gamma.
- Inflammatory bowel disease: Participants with Inflammatory Bowel Disease with a well-recognized granulomatous inflammation, but normal phagocyte function and ROS production. They have not been diagnosed with CGD.
- Other immune system disorders: Participants with other disorders such as Chediak-Higashi Syndrome, Leukocyte Adhesion Deficiency, myeloperoxidase deficiency, Hyper- IgE (Job's) Syndrome, IRAK4-deficiency, and NEMO-deficiency
- X-linked Chronic Granulomatous Disease (CGD): Participants diagnosed with X-linked CGD confirmed by DHR.

SUMMARY:
Background:

* Atherosclerosis, the arterial plaques or blockages that cause heart disease, develops in many people by the time they are in their mid-20s. The rate of atherosclerosis in patients with immune system disorders has not been well studied, but it may be very different from the general population.
* Patients with chronic granulomatous disease (CGD) produce less of a group of molecules known as free radicals, which help to fight infection and may play a role in the development of atherosclerosis. Patients with CGD may develop atherosclerosis much more slowly than people without CGD. On the other hand, carrier mothers of children with genetically-linked CGD often have problems with autoimmune problems in addition to a problem with making free radicals. Patients with other immune system disorders also have very different responses to infection, and many of them also have autoimmune-like problems that may change the risk of developing atherosclerosis.

Objectives:

- To study the prevalence of atherosclerosis in patients with immune system disorders, compared with healthy individuals.

Eligibility:

- Individuals at least 18 years of age who either have been diagnosed with an immune system disorder or are healthy volunteers.

Design:

* The active part of the study involves one or two visits to the National Institutes of Health Clinical Center for a series of imaging tests and scans.
* Participants will have the following tests during the active part of the study:
* (1) CAT scan to obtain images of the chest arteries and measure the amount of calcium in the artery walls.
* (2) Magnetic resonance imaging scan to obtain images of the coronary and carotid arteries in the chest and neck.
* (3) Electrocardiogram to provide data on current heart function.
* (4) Blood samples to provide data on heart, kidney, and immune system function.
* Participants will be contacted every 2 years in the future for up to 30 years to determine whether they have developed heart disease. Researchers will ask participants to provide contact information for two other people who may likely know how to get in touch with the participant in the future.

DETAILED DESCRIPTION:
Heart disease kills more than half a million people in the U.S. each year. Atherosclerosis, the major cause of heart disease, is thought to relate to dysregulated inflammation in the cardiovascular system and possibly results from over production of reactive oxygen species (ROS). The rate of atherosclerosis in patients with disorders of the immune system has not been well characterized but is likely to be dramatically different than that seen in the general population. Specifically, patients with Chronic Granulomatous Disease (CGD) may be protected from developing atherosclerosis due to reduced superoxide and other ROS production by phagocytic cells. We hypothesize that patients with CGD are at decreased risk of developing atherosclerosis. The primary objective of this study is to determine the prevalence of atherosclerosis and it s inflammatory characteristics in these and other patients with in-born disorders of immune function. The primary objective will be assessed using carotid studies and other imaging techniques to measure coronary artery calcium scores and the presence or absence of soft plaque. Secondary endpoints include physiologic characteristics such as blood pressure as well as circulating biomarkers associated with heart disease such as C-reactive protein and lipid profile. This study may lead to improved understanding of the pathophysiology of atherosclerosis, specifically the role of free radical stress, and could lead to novel therapies for atherosclerosis that may benefit patients with immune disorders and the general population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be identified for this protocol who are enrolled on existing protocols studying patients with disorders of the immune system who volunteer for participation and who do not have any of the listed exclusion criteria. Patients will remain enrolled on their existing protocol. Normal volunteers will be enrolled as controls on this protocol. They will be recruited through the normal volunteer office which will provide a list of volunteers including their age to allow for inclusion of controls that approximate the study population.

All patients enrolled on this protocol will be over the age of 18 and may be male or female and will be accrued without regard to religion, race or sexual orientation. They must be able to understand and sign informed consent documents and comply with study procedures that include undergoing a CT scan and an MRI scan. Patients who are unable or unwilling to complete one or more of the studies will not be excluded. The available data will be included in the appropriate analysis.

EXCLUSION CRITERIA:

For Participation in MRI-Based Studies Only:

1. Subjects with contraindication to MRI scanning. These contraindications include but are not limited to the following devices or conditions:

   1. Implanted cardiac pacemaker or defibrillator
   2. Cochlear Implants
   3. Ocular foreign body (i.e., metal shavings)
   4. Embedded shrapnel fragments
   5. Central nervous system aneurysm clips
   6. Implanted neural stimulator
   7. Medical infusion pumps
   8. Any implanted device that is incompatible with MRI
2. Patients whose medical condition is such that in the referring physicians estimation, they could not tolerate an MRI scan. Examples of medical conditions that would not be accepted would include unstable angina and dyspnea at rest.
3. Subjects with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.) or who require more than oral sedation (i.e. IV sedation) for anxiety associate with MRI studies.
4. Pregnant or lactating women are excluded from this study because excessive exposure of the developing human fetus and child to radiation and/or intravenous contrast agents can be detrimental.
5. Subjects with severe back-pain or motion disorders who will be unable to tolerate supine positioning within the MRI scanner and hold still for the duration of the examination.

   For Gadolinium-Based MRI Studies Only:
6. History of severe allergic reaction to gadolinium contrast agents despite the use of premedication with an anti-histaminic and/or corticosteroid.
7. eGFR less than 60mL/min
8. Serum creatinine greater than 3.0 mg/dl

   For Iodine-Based Contrast CT Studies Only:
9. Contraindication to the use of iodine based CT contrast agents:

   1. Serum creatinine greater than 1.4 mg/dl
   2. History of multiple myeloma
   3. Use of metformin-containing products less than 24 hours prior to contrast administration
   4. History of significant allergic reaction to CT contrast agents despite the use of premedication with an anti-histaminic and cortisone.

   For Coronary CT Angiography Only:
10. Contraindication to the use of CT contrast agents:

    1. Creatinine value greater than1.4 mg/dl
    2. History of multiple myeloma
    3. Use of metformin-containing products less than 24 hours prior to contrast administration
    4. History of significant allergic reaction to CT contrast agents despite the use of premedication with an anti-histaminic and cortisone.
11. Subjects with contraindication precluding the use of beta blockers necessary to perform the coronary CT angiography. These include:

    1. Severe, uncontrolled asthma
    2. Active bronchospasm
    3. Moderate or severe COPD
    4. 2nd or 3rd degree AV block
    5. Decompensated cardiac failure
    6. Allergy to beta blockers
    7. Systolic blood pressure less than100 mm Hg
    8. Pregnancy or nursing

    For FDG-PET:
12. Participants who are unable or unwilling to comply with the dietary modifications or physical activity restrictions prior to FDG-PET scanning will be excluded. Due to the need for dietary manipulation and maintenance of strict glycemic control we will exclude diabetic patients from our initial study sample. Blood glucose measurements before injection must be within normal limits, less than 200 mg/dl (11mmol/L).

Participation of Minors: Atherosclerosis is a disease that does not generally affect young children. This protocol involves exposure to a low dose of radiation. As radiation exposure may increase the risk of malignancy, it is prudent to avoid this in children. Therefore, patients under the age of 18 will not be considered for enrollment under this protocol.

Participation of Women: Excessive radiation exposure of the developing human fetus can be detrimental. For this reason, women of childbearing-age will have a pregnancy test prior to undergoing study procedures. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should immediately inform study staff and her primary care physician.

Pregnancy: Pregnant women are excluded from this study because excessive exposure of the developing human fetus to radiation can be detrimental.

Co-enrollment Guidelines: Co-enrollment in other trials is not restricted.

Medical Exclusions: Patients with current atrial fibrillation will not be considered for enrollment under this protocol. Patients who are medically unstable (e.g. severe sepsis, acute myocardial infarction) and/or would require active, acute medical management in order to be medically stable enough to participate in this protocol will not be enrolled.

X-linked CGD Cohort: Patients in this cohort must have X-linked CGD as demonstrated by DHR or genetic screening. Patients who have undergone bone marrow transplant may not be enrolled in this cohort for analysis. Carriers of X-linked CGD must be evaluated by DHR to determine the extent of X-inactivation (lyonization) in their neutrophils.

AutosomalRecessive CGD Cohort: Patients in this cohort must have autosomal recessive CGD (p47phox, p67phox, or p22phox deficiency) as demonstrated by DHR or genetic screening. Patients who have undergone bone marrow transplant may not be enrolled in this cohort for analysis.

Inflammatory Bowel Disease Cohort: Patients enrolled into this cohort may not have been diagnosed with CGD.

Normal Volunteer Cohort: Patients in this cohort may not have been diagnosed with CGD, Inflammatory Bowel Disease, or another primary disease of the immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified for this protocol who are enrolled on existing protocols studying patients with disorders of the immune system who volunteer for participation and who do not have any of the listed exclusion criteria. Normal volunteers will be enrolled as controls on this protocol. They will be recruited through the normal volunteer office, which will provide a list of volunteers including their age to allow for inclusion of controls that approximate the study population.All participants enrolled on this protocol will be over the age of 18 and may be male or female and will be accrued without regard to religion, race or sexual orientation.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Coronary CT angiography | September 2009- December 2024
  presence or absence of soft plaque
Coronary Artery Calcium score | September 2009- December 2024
  numerical value ranging from 0 to >1000
Coronary MRI angiography | September 2009- December 2024
  presence of absence of soft plaque
Carotid Artery Intimal Medial Thickness | September 2009- December 2024
  numerical value (in millimeters) representing the thickness of the artery and vessel wall volume
Carotid arterial FDG uptake | September 2009- December 2024
  target to background ratio of FDG activity measured by PET imaging.

SECONDARY OUTCOMES:
Circulating Markers of Cardiac Disease | September 2009- December 2024
  Lipid Profile, CRP,Myeloperoxidase analyzed for coronary artery disease risk.
Demographic Characteristics and Questionnaire Results | September 2009- December 2024
  Standard questionnaires will be used to collect information about demographics, socioeconomic and psychosocial status, medical and family history, medication use, dietary and alcohol intakes, smoking, and physical activity. Data will be analyzed using a multivariate analysis.
Physiologic Characteristics | September 2009- December 2024
  Physiologic data including blood pressure, heart rate, and pulse pressure will also be obtained. EKG will be assessed for electrocardiographic evidence of prior ischemic injury.
Circulating Markers of Inflammation or Immune Dysregulation | September 2009- December 2024
  IL-8, TNF, ESR,IFN, DHR
Cardiac MRI | September 2009- December 2024
  used to determine left ventricular wall motion and cardiac size and to determine the presence of granulomas in the ventricular wall. Results will be reported as an overall cardiac volume, left ventricular ejection fraction, the presence or absence of wall motion abnormalities, and the presence or absence of granulomas

CONTACTS AND LOCATIONS:
Overall Officials: John I Gallin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winkelstein JA, Marino MC, Johnston RB Jr, Boyle J, Curnutte J, Gallin JI, Malech HL, Holland SM, Ochs H, Quie P, Buckley RH, Foster CB, Chanock SJ, Dickler H. Chronic granulomatous disease. Report on a national registry of 368 patients. Medicine (Baltimore). 2000 May;79(3):155-69. doi: 10.1097/00005792-200005000-00003. PMID 10844935
- [Background] Lassegue B, Sorescu D, Szocs K, Yin Q, Akers M, Zhang Y, Grant SL, Lambeth JD, Griendling KK. Novel gp91(phox) homologues in vascular smooth muscle cells : nox1 mediates angiotensin II-induced superoxide formation and redox-sensitive signaling pathways. Circ Res. 2001 May 11;88(9):888-94. doi: 10.1161/hh0901.090299. PMID 11348997
- [Background] Sorescu D, Weiss D, Lassegue B, Clempus RE, Szocs K, Sorescu GP, Valppu L, Quinn MT, Lambeth JD, Vega JD, Taylor WR, Griendling KK. Superoxide production and expression of nox family proteins in human atherosclerosis. Circulation. 2002 Mar 26;105(12):1429-35. doi: 10.1161/01.cir.0000012917.74432.66. PMID 11914250
- [Derived] Sibley CT, Estwick T, Zavodni A, Huang CY, Kwan AC, Soule BP, Long Priel DA, Remaley AT, Rudman Spergel AK, Turkbey EB, Kuhns DB, Holland SM, Malech HL, Zarember KA, Bluemke DA, Gallin JI. Assessment of atherosclerosis in chronic granulomatous disease. Circulation. 2014 Dec 2;130(23):2031-9. doi: 10.1161/CIRCULATIONAHA.113.006824. Epub 2014 Sep 19. PMID 25239440
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-I-0029.html